CLINICAL TRIAL: NCT01179815
Title: Swiss Diabetes Registry - SwissDiab Study, a Prospective Cohort Study of Patients With Diabetes in Switzerland
Brief Title: Swiss Diabetes Registry - SwissDiab Study
Acronym: SwissDiab
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EKSG 01/114/L; EKSG 01/114/3B (Other: EC SG (previous number)); KEK 025/10 (Other: EC Bern (previous number))
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
Keywords: Patients with type 1 or type 2 diabetes mellitus; Monogenetic diabetes; Pancreatogenic diabetes,; Drug-induced diabetes, other forms; Cohort Studies
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and full blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with type 1 or type 2 diabetes mellitus, monogenetic diabetes, pancreatogenic diabetes, drug-induced diabetes, other forms

SUMMARY:
Currently, the estimated number of people with diabetes mellitus is approximately 387 million people worldwide. Due to population growth, urbanization, ageing and the rising prevalence of obesity the numbers of individuals with diabetes is increasing likewise. It has been shown that improving glycemic control is associated with a reduction in late complications of diabetes, such as cardiovascular and microvascular diseases. Therefore, treatment guidelines were established internationally by large and renowned associations and adopted by many countries.

For Switzerland only sparse data exist on the actual implementation of such recommendations and on patient's well-being. The Swiss Diabetes Registry - SwissDiab Study is a prospective cohort study aiming at including and collecting data of virtually all patients regularly seen and treated at the study centers (≈ 500 patients each), irrespective of type, duration of diabetes or treatment . This allows the evaluation of diabetes treatment strategies at these centers. Furthermore, risk indicators for micro- and macrovascular complications, mortality as well as costs and quality of life will be assessed. Data will be recorded through an internet-based, electronic database specifically designed for this study. At a later perspective it is planned to extend data collection to general practitioner/family doctor networks in order to include a larger and more representative sample of patients with diabetes in Switzerland.

DETAILED DESCRIPTION:
Background

Currently, approximately 387 million people worldwide are affected by Diabetes Mellitus.

Due to population growth, urbanization, ageing and the rising prevalence of obesity the numbers of individuals with diabetes will grow. The American Diabetes Association estimated the total cost of diabetes in the US in 2012 at $245 billion. The greatest share of those costs results from the treatment of diabetes-associated complications caused by prolonged hyperglycemia. There is compelling evidence that tight glycemic control and intensive treatment of other cardiovascular risk factors substantially reduce the risk of developing being also cost-effective. Our current knowledge, however, is mainly derived from intervention trials usually including strictly defined patient groups and are carried out according to meticulous study protocols. Observational studies, however, in unselected outpatient settings have revealed discrepancies between recommended treatment goals resulting from those latter studies and actual standard of care. There is a pressing need, therefore, to assess the standard of care and confirm the feasibility and effectiveness of proposed management trends in both specialty clinic and community-based cohorts.

Objective

1. With the help of an internet-based, electronic database (webspirit®, www.swissdiab.ch): to collect representative cross-sectional data from all consenting patients seen and treated at the study centers in order to evaluate the current standard of care of patients with diabetes mellitus, the distribution of micro- and macrovascular complications, the use of medications and devices as well as aspects of costs and quality of life (QoL)
2. To collect prospective data of those patients in relation to achievement of treatment goals, changes in management, risk factors for, incidence and progression of micro- and macrovascular complications, mortality as well as costs and quality of life using the same database

Methods

After obtaining informed consent, patients with diabetes mellitus willing to participate will be invited to an initial comprehensive assessment (baseline) performed at the three cantonal study centers (Inselspital Bern, Kantonsspital St. Gallen, Universitätsspital Zürich). This will be followed by face-to-face clinical/laboratory visits between one to four times yearly according to patient's individual management plans. Once a year a comprehensive review including clinical and laboratory screening for diabetes-specific complications is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of diabetes mellitus according to ADA criteria
* Informed consent

Exclusion Criteria:

* Patients with gestational diabetes mellitus, patients unable to give informed consent, legally incompetent or incapable to comply with the study terms and conditions as well as patients with significantly reduced life expectancy (<1 year) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with diabetes above age 18 are eligible for this study, irrespective of type, duration of diabetes or treatment. Diabetes will be defined according to the current diagnosis criteria suggested by the American Diabetes Association (fasting plasma glucose ≥ 7mmol/L, occasional plasma glucose ≥11.1mmol/L (plus typical symptoms), a 2hour plasma glucose of ≥11.1mmol/L after a 75g oral glucose tolerance test, or a HbA1c ≥ 6.5%), but patients under treatment with ≥2 oral hypoglycemic agents (OHA) and/or insulin in the absence of proof of a diagnosis by fasting, random plasma glucose or oral glucose tolerance test will also be included. The type of diabetes will be diagnosed clinically in most cases. In equivocal cases classification will be based on previously reported criteria with the assistance of laboratory test results.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-01; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | annually

SECONDARY OUTCOMES:
Macrovascular morbidity | annually
Microvascular morbidity | annually
Diabetes related influence on quality of Life | annually

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brändle, Prof., Principal Investigator — Div. of Endocrinology, Diabetes and Clinical Nutrition, Kantonsspital St. Gallen; Markus Laimer, PD Dr. med., Principal Investigator — Div. of Endocrinology, Diabetes and Clinical Nutrition, University Hospital Bern; Roger Lehmann, Prof., Principal Investigator — Div. of Endocrinology, Diabetes and Clin. Nutrition, University Hospital Zürich
Locations (4):
- Switzerland (4):
  - Universitätspoliklinik für Endokrinologie, Diabetologie und Klinische Ernährung, Inselspital Bern, Bern
  - Service d'endocrinologie, diabétologie et métabolisme, Lausanne
  - Klinik für Endokrinologie, Diabetologie, Osteologie und Stoffwechselerkrankungen, Kantonsspital St.Gallen, Sankt Gallen
  - Klinik für Endokrinologie, Diabetologie und Klinische Ernährung, Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No